CLINICAL TRIAL: NCT04198844
Title: The Effectiveness and Safety of Apixaban Versus Warfarin in Non-valvular Atrial Fibrillation (NVAF) Patients With the History of Osteoporosis and/or Fracture: A Nation-wide Population Based Study
Brief Title: The Effectiveness and Safety of Apixaban in NVAF Patients With History of Osteoporosis and/or Fracture: A Nation-wide Population Based Study
Status: Withdrawn | Type: Observational
Why Stopped: Interaction term analysis result was not significant and thus comparative effectiveness for primary and secondary outcomes could not be considered per protocol.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661126
Record Dates: First submitted 2019-12-02; First posted 2019-12-13 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Warfarin user
  Interventions: Drug: warfarin
- Apixaban user
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: warfarin — warfarin user
  Groups: Warfarin user
Drug: apixaban — apixaban user
  Groups: Apixaban user

SUMMARY:
Old age, less body weight and deteriorated renal function are significant clinical factors for the outcomes of atrial fibrillation- so called 'fragile'- and these are common risk factors in osteoporosis and fracture. Therefore, in real world, these risk factors and co-morbidities are commonly considered when it comes to prescribe anticoagulant in atrial fibrillation patients. Recent study even reported that comorbid atrial fibrillation in patients with osteoporosis might be associated with an increased risk of bone fracture and death after fracture. Because there have been very few data about the effectiveness/safety of anticoagulant among non-valvular atrial fibrillation with prior osteoporosis/fracture, this study is planned to provide real-world evidences for this specific type of non-valvular atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older on the index date
* Patients had ≥1 medical claim for atrial fibrillation with at least one hospitalization or at least two outpatient visits during the reference period

Exclusion Criteria:

* Patients with valvular atrial fibrillation or transient atrial fibrillation
* Having ≥ 2 types of oral anticoagulant on the index date
* who have contraindications to oral anticoagulant
* confounder factors related to the outcome (osteoporotic fractures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-valvular atrial fibrillation patients with warfarin or apixaban user
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-18 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite of ischemic stroke, hemorrhagic stroke and and systemic embolism | from index date (1st prescription date for oral anticoagulants during the intake period) to follow up period(the index date- Nov 30, 2016 or outcomes whichever comes first)
  Intake period is from July 1, 2015 to Nov 30, 2016.

SECONDARY OUTCOMES:
Major bleeding including gastrointestinal bleeding, intracranial bleeding, and other bleeding | from index date (1st prescription date for oral anticoagulants during the intake period) to follow up period (the index date- Nov 30, 2016 or outcomes whichever comes first)
  Intake period is from July 1, 2015 to Nov 30, 2016.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661126